CLINICAL TRIAL: NCT00591097
Title: Determining Normal Reference Ranges for Urinary Metabolites and Supersaturation Indices in the Pediatric Population
Brief Title: Normal Reference Ranges for Urinary Metabolites and Supersaturation Indices in Pediatric Populations
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: M-2005-1376
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: urine; pediatric; Normal urine from healthy pediatric population

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pediatric

SUMMARY:
The reported normal values used in diagnosing and treating pediatric kidney stone formers are based on adult values or historic data from small studies. Urinary supersaturation indices which are now described in the adult stone literature as more sensitive predictors of stone composition, and precise predictors of response to therapy, are not established in children. The goals of this prospective study are to redefine normal values for pediatric urinary metabolites and supersaturation indices based on samples from a large number of healthy children and to identify if a difference in urinary supersaturations in children is protective.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female children between the ages of 3 and 18, inclusive, of all races who are toilet trained and who can submit a 24-hour urine sample

Exclusion Criteria:

* Active urinary tract infection
* Known urologic anatomic abnormality
* Personal or first-degree relative family history of urolithiasis or metabolic abnormality known to lead to urinary stone development
* Renal insufficiency
* Inability to collect a 24-hour urine specimen
* Intake of medications known to alter the risk of stone development such as steroids or diuretics or vitamins or calcium supplementation exceeding recommended daily allowances
* Adherence to restrictive diet for medical reasons
* Inflammatory or absorptive bowel disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All normal, healthy volunteer children between the ages of 3 and 18, inclusive, with no personal or first relative family history of urolithiasis. Both boys and girls will be enrolled with an effort to enroll an equal number of children of all ages after toilet training.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Define normal reference ranges for urinary metabolites in the pediatric population | Assessed one time with normal urine

SECONDARY OUTCOMES:
Determine supersaturation indices in normal urine of the pediatric population | Assessed one time in normal urine

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Slaughenhoupt, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Charles Durkee, MD, Milwaukee, Wisconsin